CLINICAL TRIAL: NCT03290001
Title: The Influence of Anxiety and Depression on Survival in Nasopharyngeal Carcinoma Patients: a Prospective Observational Cohort Study
Brief Title: The Influence of Anxiety and Depression on Survival in Nasopharyngeal Carcinoma Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Deputy Director of the Department of Nasopharyngeal Carcinoma, Sun Yat-sen University
Other Study IDs: anxiety and depression
Record Dates: First submitted 2017-09-03; First posted 2017-09-21 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, observational cohort study aimed to explore the influence of anxiety and depression to long term survival in nasopharyngeal carcinoma patients.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma (NPC) is endemic in Southern China and Southeast Asia. Radiotherapy (RT) and chemotherapy are the mainstays of therapy for NPC because these tumors are biologically highly radiosensitive and chemosensitive. Anxiety and depression symptoms were common psychological symptoms around the time of cancer diagnosis and were often persistent during cancer treatment. Psychological symptoms are associated with prolonged hospital stays, lower quality of life, and worse treatment adherence among patients with cancer. Depressive symptoms have been demonstrated to predict early mortality among patients with some kinds of cancer. But among NPC patients, the influence of anxiety and depression symptoms to long term survival have not be explored. Therefore, this prospective, observational cohort study aimed to explore the influence of anxiety and depression to long term survival in NPC patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly histologically confirmed non-keratinizing nasopharyngeal carcinoma, including WHO II or III
* Age between 18-70
* Male and no pregnant female
* Patient have signed on the informed consent, and well understood the objective and procedure of this study

Exclusion Criteria:

* The presence of uncontrolled life-threatening illness
* Pregnancy or lactation
* Patient with severe medical condition

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: University hospital
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-08-20 (Actual); Primary Completion 2022-09-20 (Estimated); Study Completion 2022-09-20 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival | 3 years
  Progress-free survival is calculated from the date of registration to the date of the first progress at any site.

SECONDARY OUTCOMES:
Anxiety related measure | Baseline, completion of radiation therapy (up to 12 weeks)
  Hospital Anxiety and Depression Scale (HADS) and Hamilton Anxiety Rating Scale (HAMA) will be used during the assessment.
Distress related measure | Baseline, completion of radiation therapy (up to 12 weeks)
  Hospital Anxiety and Depression Scale (HADS) and Hamilton Depression Rating Scale (HAMD) will be used during the assessment.
Overall Survival(OS) | 3 years
  The OS was defined as the duration from the date of registration assignment to the date of death from any cause or censored at the date of the last follow-up.
Locoregional Relapse-Free Survival(LRFS) | 3 years
  The LRFS is evaluated and calculated from the date of registration until the day of first locoregional relapse or until the date of the last follow-up visit.
Distant Metastasis-Free Survival (DMFS) | 3 years
  The DMFS is evaluated and calculated from the date of registration until the day of first distant metastases or until the date of the last follow-up visit.
Complete Response (CR) | completion of radiation therapy (up to 12 weeks)
  CR assessed by independent reviewers, according to the Modified Response Evaluation Criteria in Solid Tumors (RECIST) from the National Cancer Institute (NCI). Disease response evaluated after the completion of the treatment. Complete response defined as the complete disappearance of the target and non-target lesion(s) identified at baseline after radiological evaluation by Magnetic Resonance Imaging (MRI) only.
Weight Loss | Baseline, completion of radiation therapy (up to 12 weeks)
  Weight loss was calculated as the relative percent of weight changes between weight measurement before and after the nasopharyngeal carcinoma treatment. Weight loss was calculated from the following formula:（ pro-treatment body weight - post-treatment body weight）/ pro-treatment body weight.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China